CLINICAL TRIAL: NCT02409732
Title: Photodynamic Therapy (PDT) With Levulan and Blue Light for the Treatment of Actinic Cheilitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Michael S. Chapman, Staff Physician, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D15043 28525
Record Dates: First submitted 2015-03-27; First posted 2015-04-07 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Actinic Cheilitis
Keywords: Actinic cheilitis; Photodynamic therapy; Levulan; Blue light
MeSH Terms: conditions — Actinic cheilitis | interventions — Aminolevulinic Acid; Photochemotherapy; Blue Light; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PDT (Experimental): PDT with aminolevulinic acid hydrochloride (HCl) and blue light to the affected area of the lips every six weeks for up to three treatments
  Interventions: Drug: aminolevulinic acid hydrochloride; Procedure: Photodynamic therapy with blue light

INTERVENTIONS:
Drug: aminolevulinic acid hydrochloride
  Other Names: Levulan; aminolevulinic acid HCl
Procedure: Photodynamic therapy with blue light
  Other Names: PDT with blue light; PDT

SUMMARY:
To evaluate the safety and efficacy of PDT with blue light and topical Levulan in the treatment of actinic cheilitis.

DETAILED DESCRIPTION:
The study will consist of a screening visit, up to three scheduled treatments, and two scheduled office visits. There can be a three-day window period for each scheduled visit in order to accommodate the subject's schedule and unforeseen scheduling conflicts.

1. Visit 1 (Screening): Subjects can be screened for the study up to two weeks before Visit 2 (Baseline). During screening, the study will be reviewed, written informed consent obtained, and eligibility confirmed. If applicable, the washout from prohibited medications or treatments will be determined at this visit.
2. Visit 2 (Baseline): Following signed, written informed consent and confirmation of eligibility, all subjects will have their lips photographed. Medical history, dermatologic exam, urine pregnancy test (if applicable), review of concomitant medications, clinical evaluations, and tolerability assessments will be performed at this visit. Study medication application to clean skin will be followed by a 90 minute incubation period under occlusion. Subsequently, patients will be exposed to blue light therapy for 16 minutes and 40 seconds. Post-therapy assessments will be performed afterwards, as well as education on appropriate sun protection methods.
3. Visits 3-4: Subjects will return every six weeks for up to two additional treatments. Treatment will be discontinued once the patient has achieved clinical clearance. Tolerability assessments, study medication application, blue light therapy, post-therapy assessments, and photographs will be performed.
4. Visit 5-6 (End of Study): Subjects will return 12 and 24 weeks after the last treatment for clinical evaluations, tolerability assessments, and photographs.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to understand and voluntarily sign an informed consent form
* Must be male or female ≥ 18 years of age at the time of consent
* Must be able to adhere to the study visit schedule and other protocol requirements
* Must have a diagnosis of actinic cheilitis by histopathological evaluation of biopsy specimen or clinical presentation

Exclusion Criteria:

* Inability to provide voluntarily consent or mentally incompetent
* Active herpes labialis lesions
* Subjects with any condition which places the subject at unacceptable risk if he/she were to participate in the study, or confounds the ability to interpret data from the study
* Subjects with any other skin condition that might affect the evaluation of the study disease
* Pregnant or breastfeeding female subjects
* Subjects who have used any investigational medication within one month prior to study entry
* Subjects who have been previously exposed to PDT and/or topical Levulan therapy for the treatment of actinic cheilitis
* Subjects who have used local therapy (e.g. cryotherapy) or topical treatment (e.g. 5% fluorouracil) within three months of study entry
* Subjects who have used an oral photosensitizing drug (e.g. Declomycin) within six months of study entry
* Subjects who are currently using photosensitizing agents (e.g. thiazides, tetracyclines, fluoroquinolones, phenothiazines, and sulfonamides) because of the risk of augmented photosensitivity
* Subjects who are frequently exposed to ultraviolet radiation (e.g. lifeguards, construction workers, frequent sunbed users, etc.)
* Subjects with a history of cutaneous photosensitization, porphyria, hypersensitivity to porphyrins, or photodermatosis
* Subjects with a known hypersensitivity to Levulan
* Subjects who are immunocompromised

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Chapman, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Background] Ribeiro CF, Souza FH, Jordao JM, Haendchen LC, Mesquita L, Schmitt JV, Faucz LL. Photodynamic therapy in actinic cheilitis: clinical and anatomopathological evaluation of 19 patients. An Bras Dermatol. 2012 May-Jun;87(3):418-23. doi: 10.1590/s0365-05962012000300011. PMID 22714758
- [Background] Zaiac M, Clement A. Treatment of actinic cheilitis by photodynamic therapy with 5-aminolevulinic acid and blue light activation. J Drugs Dermatol. 2011 Nov;10(11):1240-5. PMID 22052302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty four patients were screened to participate. Three men and one woman did not meet criteria to participate in the study.
Pre-assignment Details: Twenty four patients were screened to participate, but only 20 entered into the study (3 men and 1 woman screen failed). This was an open label proof of concept study and our goal was to enroll a total of 20 patients, which we achieved.
Groups:
- Photodynamic Therapy With Blue Light: Photodynamic therapy (PDT) with aminolevulinic acid hydrochloride (HCl) and blue light to the affected area of the lips every six weeks up to three treatments.
Period: Overall Study
Arm/Group | Photodynamic Therapy With Blue Light
Started | 20 (First patient consented on 4/23/15)
Completed | 14
Not Completed | 6
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Twenty four patients were screened, but only 20 were included in the study and proceeded to the baseline assessment. Nine men and 11 women RECEIVED AT LEAST ONE TREATMENT.
Arm/Group | Photodynamic Therapy With Blue Light
Number analyzed (Participants) | 20
Age, Continuous [Median (Standard Deviation); unit: years] | 65 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Income [Number; unit: participants]
  $10,000-25,000 | 1
  $26,000-50,000 | 1
  $51,000-75,000 | 4
  $76,000-100,000 | 4
  >$100,000 | 4
  Prefer not to answer | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Change in Clearance From Baseline
Description: Clearance will be estimated clinically as minimal (0%-25%), mild (26%-50%), moderate (51%-75%), good (76%-99%), or complete (100%). Results will also be evaluated by comparing photographs before and immediately after treatments, and 12 and 24 weeks after the last treatment.
Time Frame: Visit 2 (Baseline) to Visit 5 or 6 (Week 24 or 36)
Population: Twenty patients were enrolled into the study. Please see baseline characteristics to understand the patient demographic.
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy With Blue Light
Number analyzed (Participants) | 20
Participants
  0% improvement at V6 (week 36) | 1
  50% improvement at V6 (week 36) | 1
  75% improvement at V6 (week 36) | 9
  100% % improvement at V6 (week 36) | 4
  Discontinued/Withdrew/Lost to follow up | 5

2. Secondary Outcome: Average Change in Participant Reported Pain
Description: Subject reported pain before, during and after blue light illumination was documented using a Visual Analogue Scale (VAS) from 0 (no pain) to 10 (worst pain imaginable). The maximum change in pain is 10 for each occurrence (pain before compared to during treatment and pain during compared to after treatment). This is multiplied by the number of subjects and then divided by the number of treatments to generate the range. The summation of the change between subject reported pain prior to compared to during blue light treatment was divided by the total number of treatments to obtain the average value. The summation of the change between subject reported pain during compared to after blue light treatment was divided by the total number of treatments to obtain the average value.
Time Frame: Baseline to Week 36
Population: Twenty participants completed 50 treatments and the change in local skin reaction (pre-treatment, during treatment and post-treatment) was evaluated at each visit.
  Number of Patients by Number of Treatments received:
  One Treatment: 4 Two Treatments :2 Three Treatments:14
Measure: Mean (Full Range); unit: units on a scale
Units Other Than Participants: Treatment visits
Arm/Group | Photodynamic Therapy With Blue Light
Number analyzed (Participants) | 20
Number analyzed (Treatment visits) | 50
units on a scale
  Avg change of pain prior to tx to during tx | 2.86 [-4 to 4]
  Avg change of pain during tx to after tx | -0.76 [-4 to 4]

3. Secondary Outcome: Average Change in Local Skin Reactions to Blue Light Treatment
Description: Assessments of swelling, erythema, and flaking/scaling were conducted after each treatment and two days post-treatment using a five-point ordinal scale (0: none to 4: severe). The average change in swelling, erythema and flaking/scaling after each treatment and two days post treatment were divided by the 50 total treatments to obtain the average value.
Time Frame: Baseline to Week 36
Population: Twenty participants completed 50 treatments and the change in local skin reaction (pre-treatment, during treatment and post-treatment) was evaluated at each visit.
Measure: Mean (Full Range); unit: units on a scale
Units Other Than Participants: Treatment visits
Arm/Group | Photodynamic Therapy With Blue Light
Number analyzed (Participants) | 20
Number analyzed (Treatment visits) | 50
units on a scale
  Swelling | 0.72 [-1 to 3]
  Erythema | 0.58 [-2 to 3]
  Flaking/Scaling (Skin Dryness) | 1.82 [0 to 4]

4. Secondary Outcome: The Number of Participants Who Developed a Local Skin Reaction to Blue Light Treatment: Vesiculation/Pustulation, Erosion/Ulceration, Crusting and Hyperpigmentation
Description: Assessments of vesiculation/pustulation, erosion/ulceration, and crusting were conducted immediately after each blue light treatment using a five-point ordinal scale (0: none to 4: severe). The presence or absence of hyperpigmentation in the treatment area was also documented after each treatment visit. The total number of participants who developed a local skin reaction is documented.
Time Frame: Baseline to Week 36
Population: as for outcome 3
Measure: Number; unit: participants
Units Other Than Participants: Treatment visits
Arm/Group | Photodynamic Therapy With Blue Light
Number analyzed (Participants) | 20
Number analyzed (Treatment visits) | 50
participants
  Vesiculation/Pustulation | 2
  Erosion/Ulceration | 0
  Crusting | 4
  Hyperpigmentation | 1

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Evaluation of any reported local or systemic events outside the treatment area and other than those specified under local skin reactions or PDT reactions.
Time Frame: Baseline to Week 36
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy With Blue Light
Number analyzed (Participants) | 20
Participants
  Upper respiratory infection (URI) | 1
  Lesion on mid chest | 1
  Red spots | 1
  Bleeding esophageal ulcer | 1

ADVERSE EVENTS:
Time Frame: Visits 2 (Baseline), Visits 3 (week 6), and Visit 4 (week 12), Visit 5 (week 24), Visit 6 (week 36)
Arm/Group | Photodynamic Therapy With Blue Light
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 3/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Photodynamic Therapy With Blue Light (N=20)
Bleeding esophageal ulcer (Gastrointestinal disorders) | 1 (1) — Bleeding esophageal ulcer requiring inpatient hospitalization during the study treatment. This was deemed unrelated to the study treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Photodynamic Therapy With Blue Light (N=20)
URI (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Swelling of right hand (Skin and subcutaneous tissue disorders) | 1 (1) — Patient underwent mohs surgery on the right hand. This adverse event was not related to the study treatment.
Red spots (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT02409732/Prot_SAP_000.pdf